CLINICAL TRIAL: NCT01965821
Title: Impact of Mallinckrodt Electronic Device on Continuous Control of Tracheal Cuff Pressure
Acronym: RCPBALSTAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2012_41; 2013 A00225 40 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2013-10-16; First posted 2013-10-18 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2017-03

CONDITIONS: Critical Illness
Keywords: tracheal cuff pressure; continuous control; microaspiration
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continuous control of Pcuff followed by manual control (Other): Patients receive continuous control of cuff pressure with Mallinckrodt electronic device for 24h, followed by discontinuous control (every 8 hours) with a manual manometer for 24h.
  Interventions: Device: Continuous control of Pcuff followed by manual control
- Manual control of Pcuff followed by continuous control (Other): Patients receive the reverse sequence (manual control followed by continuous control of Pcuff)
  Interventions: Device: Manual control of Pcuff followed by continuous control

INTERVENTIONS:
Device: Continuous control of Pcuff followed by manual control — continuous control of tracheal cuff pressure using an electronic device for 24 h followed by manual control of cuff pressure using a manometer
  Arms: Continuous control of Pcuff followed by manual control
Device: Manual control of Pcuff followed by continuous control — 24 h of manual control using a manometer followed by 24 h of continuous control using an electronic device
  Arms: Manual control of Pcuff followed by continuous control

SUMMARY:
Despite intermittent control of tracheal cuff pressure using a manual manometer, cuff underinflations and overinflations frequently occur in critically ill patients, resulting in increased risk for microaspiration and tracheal ischemic lesions. The aim of this study is to determine the efficiency of Mallinckrodt electronic device (Mallinckrodt electronic cuff pressure controller, VBM Medizintechnik GmbH, Sulz aN) in continuous control of tracheal cuff pressure.

ELIGIBILITY:
Inclusion Criteria: :

* Patients intubated in the ICU with a high volume / low pressure PVC-cuffed tracheal tube
* Predicted duration of mechanical ventilation > or = 48h
* Age > or = 18 years
* signed informed consent

Exclusion Criteria:

* Contraindication for semirecumbent position
* Contraindication for enteral nutrition
* Pregnancy
* refuse to participate to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
percentage of recording time spent with cuff overinflation or underinflation | 48 hours
  Continuous recording of cuff pressure will be performed during 2 24-h periods (with or without Mallinckrodt device)

SECONDARY OUTCOMES:
Impact of Mallinckrodt electronic device on microaspiration of gastric contents, documented by pepsin levels in tracheal aspirates | 48 hours
  Pepsin will be quantitatively measured in tracheal aspirates of all patients during the 2 24-h periods (with or without Mallinckrodt device)

CONTACTS AND LOCATIONS:
Overall Officials: Saad NSEIR, MD, Principal Investigator — University Hospital of Lille
Locations (1):
- ICU, Salengro Hospital, University Hospital of Lille, Lille, Nord, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rouze A, De Jonckheere J, Zerimech F, Labreuche J, Parmentier-Decrucq E, Voisin B, Jaillette E, Maboudou P, Balduyck M, Nseir S. Efficiency of an electronic device in controlling tracheal cuff pressure in critically ill patients: a randomized controlled crossover study. Ann Intensive Care. 2016 Dec;6(1):93. doi: 10.1186/s13613-016-0200-2. Epub 2016 Oct 4. PMID 27704488